CLINICAL TRIAL: NCT01900457
Title: Vestibular and Multisensory Influence on Bodily and Spatial Representations. Behavioral and Electrophysiological Investigations in Vestibular-defective Patients and Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-A01221-40; 2013-18 (Other: AP HM)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Vestibular-defective Patients
MeSH Terms: interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volunteer healthy (Active Comparator): healthy volunteers
  Interventions: Other: approaches from psychophysics
- patients (Experimental): vestibular defective patients
  Interventions: Other: electromyography; Other: electroencephalography

INTERVENTIONS:
Other: electromyography
  Arms: patients
Other: electroencephalography
  Arms: patients
Other: approaches from psychophysics
  Arms: Volunteer healthy

SUMMARY:
The present project aims at describing how vestibular signals contribute to the multisensory mechanisms of bodily self-consciousness.

There is a large body of data regarding the sensory and neural mechanisms of self-consciousness, but most studies have so far demonstrated the contribution of visual, tactile and proprioceptive signals to bodily self-consciousness. Thus, most studies have neglected the contribution of the vestibular system, a major sensory system for spatial and bodily representations. The vestibular system is sensitive to head motions in space and head inclinations with respect to gravity and it should therefore contribute significantly to several bodily experiences. This contribution should be put under neuroscientific scrutiny. We believe that the current neuroscientific models of bodily self-consciousness will be incomplete until they incorporate the contribution of vestibular signals.

The present project specifically aims at testing the hypothesis according to which vestibular signals significantly influence bodily self-consciousness, in particular first-person and third-person perspective taking and the internal body models (i.e. the body schema and body image). The present project also aims at describing how cortical vestibular processing is modified during experimental changes of perspective taking and viewpoint. In addition, the present project will describe whether vestibular disorders change performances in third-person perspective taking tasks and modify internal body models. This should help understanding bodily symptoms in vestibular-defective patients. To this end, we will combine approaches from psychophysics and electrophysiology (electromyography, electroencephalography) in healthy volunteers and behavioral approached in patients with vestibular disorders.

These studies should further the understanding of how the brain processes vestibular signals, which is to date poorly understood. In addition, the outcome of the present project should help understanding the multiple and complex symptoms reported by patients with vestibular diseases, and should therefore improve their treatment.

ELIGIBILITY:
Inclusion Criteria:

* men(people) or women from 18 to 65 years old
* patients having benefited from a surgical operation (neurotomie vestibulaire unilateral) within the framework of a disease of invalidating Ménière or a neurinome of the accoustique, or patients with an acute(sharp) infringement(achievement) of the system vestibulaire.

Exclusion Criteria:

The patients suffering from an additional hurt of the central nervous system,

* the patients suffering from driving infringements(achievements),
* the subjects having neurological histories (other than those led(inferred) by the disorders(confusions) vestibulaires) or psychiatric,
* the vulnerable persons aimed by articles L. 1121-5, L. 1121-6 and L. 1121-8,
* the persons unfit of the reading and the writing of French not allowing the understanding of the note of information and the form of consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
vestibular signals | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France